CLINICAL TRIAL: NCT05368857
Title: A Mechanistic Study to Evaluate Impact of Subcutaneous Implants of Afamelanotide on Ultraviolet Radiation-induced DNA Damage and DNA Repair Capacity in Healthy Volunteers With Skin Types I-III
Brief Title: DNA Repair Capacity of Afamelanotide on Ultraviolet Radiation-induced DNA Damage in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clinuvel (UK) Ltd. (Industry)
Responsible Party: Sponsor
Organization: Clinuvel Pharmaceuticals Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CUV151
Record Dates: First submitted 2022-04-21; First posted 2022-05-10 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Afamelanotide Evaluated as Skin DNA Repair Therapy in Healthy Volunteers
MeSH Terms: interventions — afamelanotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Afamelanotide (Experimental)
  Interventions: Drug: Afamelanotide

INTERVENTIONS:
Drug: Afamelanotide — Up to 10 adult healthy volunteers will be enrolled in this study in which small areas of their skin will be exposed to UVR and skin samples taken. UV-induced DNA damage and repair will be analysed.

SUMMARY:
This mechanistic study's aim is to assess the DNA damage repair capabilities of afamelanotide in healthy volunteers with skin type I-III following exposure to ultraviolet radiation (UVR)-induced DNA damage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers (aged 18-45) with Fitzpatrick skin types I, II or III.
* Written informed consent obtained from volunteers prior to study-start.

Exclusion Criteria:

* Female who is pregnant or lactating.
* Females of child-bearing potential not using adequate contraceptive measures or a lifestyle excluding pregnancy.
* Sexually active man with a partner of child-bearing potential who is not using adequate contraceptive measures.
* Any significant illness during the four weeks before the study screening period.
* Taking known photosensitisers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in UV photoproduct levels in UVR-exposed skin. | From Baseline to Day 28
  Analysis of UV photoproducts from skin samples.
Change in rate of UV photoproduct repair in UVR-exposed skin. | From Baseline to Day 28.
  Analysis of UV photoproduct repair mechanisms from skin samples.

SECONDARY OUTCOMES:
Change in UV-induced DNA damage and repair markers. | From Baseline to Day 28
  Analysis of UV photoproducts and DNA repair mechanisms from skin samples.
Change in Minimal Erythema Dose (MED). | From Baseline to Day 28
  Minimal erythema dose (MED) is the lowest dose of UV light that causes reddening of the skin.
Change in UVR-erythema dose-response. | From Baseline to Day 28
  UVR erythema dose response measured with a non-invasive quantitative skin reflectance measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- CLINUVEL Investigational Site, Clinuvel Investigational Site, United Kingdom